CLINICAL TRIAL: NCT02666573
Title: Effects of Photodynamic Therapy on Clinical and Immunological Parameters in a Group of Periodontal Patients Undergoing Supportive Periodontal Therapy
Brief Title: Photodynamic Therapy During Supportive Periodontal Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Goh Xian Jun Edwin, Periodontology Resident, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R-221-000-044-597
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Periodontal Diseases; Chronic Periodontitis; Periodontal Attachment Loss
Keywords: drug therapy; Photosensitizing Agents; therapeutic use
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis; Periodontal Attachment Loss | interventions — Tooth Exfoliation; Root Planing

ARMS (2):
- Photodynamic therapy protocol (Experimental): In addition to scaling and root debridement, test sites received PDT according to manufacturer's instructions.
  Interventions: Device: Fotosan 630, CMS Dental, Copenhagen, Denmark
- SRP (Other): Scaling and root debridement of the residual pockets were performed using ultrasonic device and hand curettes until root surfaces felt hard and smooth. The sites were then polished using rubber cup and prophylaxis paste.
  Interventions: Other: Scaling and root planing

INTERVENTIONS:
Device: Fotosan 630, CMS Dental, Copenhagen, Denmark — The PDT system consists of a hand-held rechargeable light-emitting diode (LED) light source (Fotosan® 630 device, CMS Dental, Copenhagen, Denmark) and 0.1 mg/mL toluidine blue photosensitiser. The LED light source has a wavelength between 620 to 640 nm and peak of 630 nm and a power density between 2000 to 4000 mW/cm2.
  Arms: Photodynamic therapy protocol
Other: Scaling and root planing — Scaling and root debridement of the residual pockets were performed using ultrasonic device and hand curettes until root surfaces felt hard and smooth. The sites were then polished using rubber cup and prophylaxis paste.
  Arms: SRP

SUMMARY:
27 subjects on SPT, each with at least two residual pockets ≥5mm, were recruited for this randomised, split-mouth controlled trial, providing a total of 72 sites. At baseline, probing pocket depth (PPD), recession, clinical attachment level (CAL), plaque and bleeding on probing (BOP) of all sites were examined. Gingival crevicular fluid (GCF) were collected to determine level of cytokines IL-1β, -6, -8, TNF-α and MMP-8 via ELISA. Control sites received subgingival instrumentation and rubber cup polishing with pumice. In addition test sites received a single application of PDT using Fotosan® and photosensitizer consisting of toludine blue O solution. The subjects were recalled three and six months later and re-examined. Site level analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health with no systemic diseases causing manifestation of periodontal diseases
2. Age ≥ 21 years
3. History of chronic periodontitis
4. At least two residual PPD ≥ 5 mm with or without bleeding on probing
5. Compliant with recalls, i.e. last SPT visit at most 6 months before start of trial
6. Able to give written informed consent

Exclusion Criteria:

1. Pregnant or lactating females
2. Local or systemic antibiotics intake in the past 3 months
3. Systemic conditions which could affect progression of periodontitis
4. Long term use of NSAIDs or immunosuppressive medications
5. Participation in other clinical trials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in percentage change in probing pocket depth | 6 months

SECONDARY OUTCOMES:
Bleeding on probing | 6 months
Clinical attachment level | 6 months
Recession | 6 months
Cytokines level | 6 months